CLINICAL TRIAL: NCT01377584
Title: COMMENCE Study: COMMunication and Education for the New CPAP Experience
Brief Title: COMMunication and Education for the New CPAP Experience
Acronym: COMMENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Faith Luyster, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 1K23HL105887-01A1 (NIH)
Record Dates: First submitted 2011-06-17; First posted 2011-06-21 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Continuous Positive Airway Pressure; Patient Compliance; Intervention Studies; Spouses
MeSH Terms: conditions — Sleep Apnea, Obstructive; Patient Compliance | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Patients in the Couple-oriented intervention (Experimental): Patients randomly assigned to the couple-oriented (CO) group will attend two face to face sessions with their partner and participate in an individual telephone follow-up session.
  Interventions: Behavioral: Couple-oriented intervention; Device: Continuous positive airway pressure (CPAP)
- Patients in Usual Care (Other): Patients will not attend any intervention sessions.
  Interventions: Device: Continuous positive airway pressure (CPAP)
- Patients in the Patient-oriented intervention (Experimental): Patients randomly assigned to the patient-oriented (PT) group will attend two face to face sessions and participate in a telephone follow-up session.
  Interventions: Behavioral: Patient-oriented intervention; Device: Continuous positive airway pressure (CPAP)
- Partners in the Couple-oriented intervention (Experimental): Partners randomly assigned to the couple-oriented (CO) group will attend two face to face sessions with the patient and participate in an individual telephone follow-up session.
  Interventions: Behavioral: Couple-oriented intervention
- Partners in Usual Care (Other): Partners will not attend any intervention sessions.
  Interventions: Other: No intervention
- Partners in the Patient-oriented intervention (Experimental): Partners randomly assigned to the patient-oriented (PT) group will not attend any intervention sessions.
  Interventions: Behavioral: Patient-oriented intervention

INTERVENTIONS:
Behavioral: Couple-oriented intervention — The first session will occur before the patient receives his/her CPAP and will last approximately 2 hours. This session will provide the couple with education on sleep apnea and CPAP and information on different types of PAP therapy and cleaning procedures, explore patient's concerns about starting CPAP treatment, and provide a goal setting exercise. The second face to face session will occur one week after the patient receives his/her CPAP and will last approximately one and a half hours. The second session will provide the couple with information on CPAP usage and pre- and post-treatment AHI, explore barriers to CPAP use and benefits of CPAP use, and provide a goal setting exercise. The individual telephone follow-up sessions will occur two weeks after the patient has received his/her CPAP and will last approximately 20 minutes. This session will review CPAP usage and explore barriers and facilitators of CPAP use.
  Arms: Partners in the Couple-oriented intervention; Patients in the Couple-oriented intervention
Behavioral: Patient-oriented intervention — The first session will occur before the patient receives his/her CPAP and will last approximately one and a half hours. This session will provide the patient with education on sleep apnea and CPAP and information on different types of PAP therapy and cleaning procedures, explore patient's concerns about starting CPAP treatment, and provide a goal setting exercise. The second face to face session will occur one week after the patient receives his/her CPAP and will last approximately 45 minutes. The second session will provide information on CPAP usage and pre- and post-treatment AHI, explore barriers to CPAP use and benefits of CPAP use, and provide a goal setting exercise. The telephone follow-up session will occur two weeks after the patient has received his/her CPAP and will last approximately 20 minutes. This session will review CPAP usage and explore barriers and facilitators of CPAP use.
  Arms: Partners in the Patient-oriented intervention; Patients in the Patient-oriented intervention
Device: Continuous positive airway pressure (CPAP) — CPAP is treatment for obstructive sleep apnea. CPAP therapy keeps the airway open during the night by providing a stream of air through a mask that is worn while sleeping.
  Arms: Patients in Usual Care; Patients in the Couple-oriented intervention; Patients in the Patient-oriented intervention
Other: No intervention — No intervention will be received.
  Arms: Partners in Usual Care

SUMMARY:
The purpose of this research study is to examine the effect of a couple-oriented education and support intervention on patient- and partner -reported outcomes (positive airway pressure (PAP) adherence) in patients newly diagnosed with obstructive sleep apnea (OSA).

DETAILED DESCRIPTION:
Continuous positive airway pressure (CPAP) therapy is an effective treatment for obstructive sleep apnea (OSA), but adherence is poor. CPAP adherence interventions to date have been met with limited success. Intervention strategies would be optimized by added support for patients and alternative strategies for intervention delivery. Significant others (SO) are likely to exert positive and negative effects on the patient's adoption and use of positive airway pressure (PAP) therapy and are frequently described as the greatest source of social support for patients with chronic illness. Beginning the intervention before PAP initiation would capitalize on the teachable moment shortly following diagnosis when education and social support may be most essential. The aims of the research plan are to examine the effects of a couple-oriented education and support intervention on patient- and partner-reported outcomes as compared to a patient-oriented education and support intervention and usual care and to examine the relationship between PAP adherence and patients' and partners' sleep quality and daytime functioning. Patients in the pilot study will be randomized to the couple-oriented intervention, patient-oriented intervention, or standard clinical care group.

ELIGIBILITY:
Inclusion Criteria:

Patient:

* Age is 21 years of age and older
* Have spouse or partner
* Polysomnographically (PSG) diagnosed OSA (AHI ≥ 5)
* Choice of continuous positive airway pressure (CPAP) as preferred treatment

Partner:

* Age is 18 years of age and older
* Have spouse or partner who has been diagnosed with OSA and has chosen CPAP as preferred treatment

Exclusion Criteria:

Patient:

* AHI < 5 on the diagnostic PSG
* Have a spouse or partner with OSA diagnosis and on OSA treatment
* Past treatment for OSA
* Diagnosis of a sleep disorder other than OSA that cause arousals from sleep (e.g., central sleep apnea, periodic limb movement disorder, insomnia)
* Diagnosis of a serious medical condition (e.g., end stage renal failure, severe chronic obstructive lung disease, severe asthma)
* History of or current diagnosis of a major psychiatric illness except depression (e.g., schizophrenia, bipolar disorder) partner:
* Have been diagnosed with OSA and using CPAP

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faith S Luyster, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Cartwright R. Sleeping together: a pilot study of the effects of shared sleeping on adherence to CPAP treatment in obstructive sleep apnea. J Clin Sleep Med. 2008 Apr 15;4(2):123-7. PMID 18468310
- [Background] Hoy CJ, Vennelle M, Kingshott RN, Engleman HM, Douglas NJ. Can intensive support improve continuous positive airway pressure use in patients with the sleep apnea/hypopnea syndrome? Am J Respir Crit Care Med. 1999 Apr;159(4 Pt 1):1096-100. doi: 10.1164/ajrccm.159.4.9808008. PMID 10194151
- [Background] Baron KG, Smith TW, Berg CA, Czajkowski LA, Gunn H, Jones CR. Spousal involvement in CPAP adherence among patients with obstructive sleep apnea. Sleep Breath. 2011 Sep;15(3):525-34. doi: 10.1007/s11325-010-0374-z. Epub 2010 Jun 15. PMID 20549372
- [Background] Baron KG, Smith TW, Czajkowski LA, Gunn HE, Jones CR. Relationship quality and CPAP adherence in patients with obstructive sleep apnea. Behav Sleep Med. 2009;7(1):22-36. doi: 10.1080/15402000802577751. PMID 19116799
- [Background] Bazzano LA, Khan Z, Reynolds K, He J. Effect of nocturnal nasal continuous positive airway pressure on blood pressure in obstructive sleep apnea. Hypertension. 2007 Aug;50(2):417-23. doi: 10.1161/HYPERTENSIONAHA.106.085175. Epub 2007 Jun 4. PMID 17548722
- [Background] Campos-Rodriguez F, Pena-Grinan N, Reyes-Nunez N, De la Cruz-Moron I, Perez-Ronchel J, De la Vega-Gallardo F, Fernandez-Palacin A. Mortality in obstructive sleep apnea-hypopnea patients treated with positive airway pressure. Chest. 2005 Aug;128(2):624-33. doi: 10.1378/chest.128.2.624. PMID 16100147
- [Background] Aloia MS, Arnedt JT, Riggs RL, Hecht J, Borrelli B. Clinical management of poor adherence to CPAP: motivational enhancement. Behav Sleep Med. 2004;2(4):205-22. doi: 10.1207/s15402010bsm0204_3. PMID 15600056
- [Background] Sparrow D, Aloia M, Demolles DA, Gottlieb DJ. A telemedicine intervention to improve adherence to continuous positive airway pressure: a randomised controlled trial. Thorax. 2010 Dec;65(12):1061-6. doi: 10.1136/thx.2009.133215. Epub 2010 Sep 29. PMID 20880872
- [Background] Aloia MS, Di Dio L, Ilniczky N, Perlis ML, Greenblatt DW, Giles DE. Improving compliance with nasal CPAP and vigilance in older adults with OAHS. Sleep Breath. 2001;5(1):13-21. doi: 10.1007/s11325-001-0013-9. PMID 11868136
- [Background] Aloia MS, Arnedt JT, Stepnowsky C, Hecht J, Borrelli B. Predicting treatment adherence in obstructive sleep apnea using principles of behavior change. J Clin Sleep Med. 2005 Oct 15;1(4):346-53. PMID 17564399
- [Background] Aloia MS, Arnedt JT, Stanchina M, Millman RP. How early in treatment is PAP adherence established? Revisiting night-to-night variability. Behav Sleep Med. 2007;5(3):229-40. doi: 10.1080/15402000701264005. PMID 17680733
- [Background] Weaver TE, Maislin G, Dinges DF, Bloxham T, George CF, Greenberg H, Kader G, Mahowald M, Younger J, Pack AI. Relationship between hours of CPAP use and achieving normal levels of sleepiness and daily functioning. Sleep. 2007 Jun;30(6):711-9. doi: 10.1093/sleep/30.6.711. PMID 17580592
- [Background] Weaver TE, Kribbs NB, Pack AI, Kline LR, Chugh DK, Maislin G, Smith PL, Schwartz AR, Schubert NM, Gillen KA, Dinges DF. Night-to-night variability in CPAP use over the first three months of treatment. Sleep. 1997 Apr;20(4):278-83. doi: 10.1093/sleep/20.4.278. PMID 9231953
- [Background] Berg CA, Upchurch R. A developmental-contextual model of couples coping with chronic illness across the adult life span. Psychol Bull. 2007 Nov;133(6):920-54. doi: 10.1037/0033-2909.133.6.920. PMID 17967089
- [Background] Engleman HM, Martin SE, Douglas NJ. Compliance with CPAP therapy in patients with the sleep apnoea/hypopnoea syndrome. Thorax. 1994 Mar;49(3):263-6. doi: 10.1136/thx.49.3.263. PMID 8202884
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Weaver TE, Laizner AM, Evans LK, Maislin G, Chugh DK, Lyon K, Smith PL, Schwartz AR, Redline S, Pack AI, Dinges DF. An instrument to measure functional status outcomes for disorders of excessive sleepiness. Sleep. 1997 Oct;20(10):835-43. PMID 9415942
- [Background] Stepnowsky CJ Jr, Marler MR, Ancoli-Israel S. Determinants of nasal CPAP compliance. Sleep Med. 2002 May;3(3):239-47. doi: 10.1016/s1389-9457(01)00162-9. PMID 14592213
- [Background] Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Med Care. 1986 Jan;24(1):67-74. doi: 10.1097/00005650-198601000-00007. PMID 3945130
- [Background] Pierce GR, Sarason IG, Sarason BR. General and relationship-based perceptions of social support: are two constructs better than one? J Pers Soc Psychol. 1991 Dec;61(6):1028-39. doi: 10.1037//0022-3514.61.6.1028. PMID 1774625

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients in the Couple-oriented Intervention: Patients randomly assigned to the couple-oriented (CO) group will attend two face to face sessions and participate in an individual telephone follow-up session.
  Couple-oriented intervention: The first session will occur before the patient receives his/her CPAP. This session will provide the couple with education on sleep apnea and CPAP, demonstration of PAP equipment, explore patient's concerns about starting CPAP treatment, and provide a goal setting exercise. The second face to face session will occur one week after the patient receives his/her CPAP. The second session will provide the couple with information on CPAP usage and pre- and post-treatment AHI, explore barriers to CPAP use and benefits of CPAP use, and provide a goal setting exercise. The individual telephone follow-up sessions will occur two weeks after the patient has received his/her CPAP. This session will review CPAP usage and explore barriers and facilitators of CPAP use.
- Patients in the Patient-oriented Intervention: Patients randomly assigned to the patient-oriented (PT) group will attend two face to face sessions and participate in a telephone follow-up session.
  Patient-oriented intervention: The first session will occur before the patient receives his/her CPAP. This session will provide the patient with education on sleep apnea and CPAP, demonstration of PAP equipment, explore patient's concerns about starting CPAP treatment, and provide a goal setting exercise. The second face to face session will occur one week after the patient receives his/her CPAP. The second session will provide the patient with information on CPAP usage and pre- and post-treatment AHI, explore barriers to CPAP use and benefits of CPAP use, and provide a goal setting exercise. The telephone follow-up sessions will occur two weeks after the patient has received his/her CPAP. This session will review CPAP usage and explore barriers and facilitators of CPAP use.
Period: Overall Study
Arm/Group | Patients in the Couple-oriented Intervention | Partners in the Couple-oriented Intervention | Patients in the Patient-oriented Intervention | Partners in the Patient-oriented Intervention | Patients in Usual Care | Partners in Usual Care
Started | 8 | 8 | 10 | 10 | 12 | 12
Completed | 5 | 5 | 6 | 6 | 9 | 9
Not Completed | 3 | 3 | 4 | 4 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients in the Couple-oriented Intervention | Partners in the Couple-oriented Intervention | Patients in the Patient-oriented Intervention | Partners in the Patient-oriented Intervention | Patients in Usual Care | Partners in Usual Care | Total
Number analyzed (Participants) | 5 | 5 | 6 | 6 | 9 | 9 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (14) | 43 (3) | 50 (11) | 54 (14) | 54 (7) | 54 (7) | 52 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 2 | 3 | 3 | 6 | 19
  Male | 4 | 1 | 4 | 3 | 6 | 3 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 3 | 3 | 4 | 12
  White | 5 | 5 | 3 | 2 | 5 | 3 | 23
  More than one race | 0 | 0 | 1 | 1 | 1 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Apnea-Hypopnea Index [Mean (Standard Deviation); unit: Events per hour of sleep] — Apnea-Hypopnea Index is a measure of the total number of apnea and hypopnea events per hour of sleep.
  Events per hour of sleep | 40 (40) | NA (NA) — Data not collected for partners. | 30 (32) | NA (NA) — Data not collected for partners. | 40 (28) | NA (NA) — Data not collected for partners. | 37 (31)

OUTCOME MEASURES:

1. Primary Outcome: Daytime Sleepiness
Description: The Epworth Sleepiness Scale is an 8-item questionnaire that assesses daytime sleepiness.Total scores range from 0 to 24. A score of > 10 indicates excessive daytime sleepiness.
Time Frame: baseline and 3 months after CPAP initiation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients in the Couple-oriented Intervention | Partners in the Couple-oriented Intervention | Patients in the Patient-oriented Intervention | Partners in the Patient-oriented Intervention | Patients in Usual Care | Partners in Usual Care
Number analyzed (Participants) | 5 | 5 | 6 | 6 | 9 | 9
units on a scale
  Baseline | 9.0 (6.9) | 3.8 (1.9) | 6.8 (6.8) | 6.5 (4.6) | 10.8 (5.9) | 7.3 (5.2)
  3 month follow-up | 4.2 (0.8) | 1.5 (2.5) | 3.3 (2.1) | 6.9 (4.5) | 6.4 (4.8) | 4.7 (3.4)
  Change from Baseline to 3 months | -4.8 (0.8) | -1.8 (1.0) | -3.5 (6.7) | 0.4 (4.2) | -4.3 (4.6) | -2.7 (3.1)
Statistical Analysis 1: Comparison: Patients in the Couple-oriented Intervention; Test type: Other; Effect size = -0.51
Statistical Analysis 2: Comparison: Patients in the Patient-oriented Intervention; Test type: Other; Effect size = -0.42
Statistical Analysis 3: Comparison: Patients in Usual Care; Test type: Other; Effect size = -0.82
Statistical Analysis 4: Comparison: Partners in the Couple-oriented Intervention; Test type: Other; Effect size = -1.31
Statistical Analysis 5: Comparison: Partners in the Patient-oriented Intervention; Test type: Other; Effect size = -0.08
Statistical Analysis 6: Comparison: Partners in Usual Care; Test type: Other; Effect size = -0.77

2. Primary Outcome: Sleep-related Functional Outcomes
Description: The Functional Outcomes of Sleep Questionnaire-10 is 10-item questionnaire assesses the impact of sleep disorders of excessive sleepiness on multiple activities of everyday living. Scores for five domains of functioning (e.g., activity, vigilance, intimacy and sexual relationships, general productivity, and social outcome) are obtained. Each domain score ranges from 1 to 4 (1 indicating more difficulty). The total score is derived by calculating the mean of the domain scores and multiplying by five. The total score ranges from 5 to 20, with higher scores indicating greater functioning.
Time Frame: baseline and 3 months after CPAP initiation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients in the Couple-oriented Intervention | Partners in the Couple-oriented Intervention | Patients in the Patient-oriented Intervention | Partners in the Patient-oriented Intervention | Patients in Usual Care | Partners in Usual Care
Number analyzed (Participants) | 5 | 5 | 6 | 6 | 9 | 9
units on a scale
  Baseline | 16.6 (2.6) | 16.7 (2.6) | 17.2 (3.3) | 16.9 (3.9) | 15.6 (4.3) | 17.3 (2.4)
  3 month follow-up | 17.9 (0.9) | 18.2 (2.1) | 19.1 (1.5) | 17.3 (2.9) | 17.7 (2.8) | 18.0 (1.6)
  Change from Baseline to 3 months | 2.1 (3.0) | 1.5 (0.7) | 1.9 (3.7) | 0.0 (1.8) | 2.1 (3.3) | 0.8 (1.1)
Statistical Analysis 1: Comparison: Patients in the Couple-oriented Intervention; Test type: Other; Effect size = 0.51
Statistical Analysis 2: Comparison: Patients in the Patient-oriented Intervention; Test type: Other; Effect size = 0.41
Statistical Analysis 3: Comparison: Patients in Usual Care; Test type: Other; Effect size = 0.57
Statistical Analysis 4: Comparison: Partners in the Couple-oriented Intervention; Test type: Other; Effect size = 1.54
Statistical Analysis 5: Comparison: Partners in the Patient-oriented Intervention; Test type: Other; Effect size = 0.00
Statistical Analysis 6: Comparison: Partners in Usual Care; Test type: Other; Effect size = 0.65

3. Primary Outcome: Sleep Quality
Description: The Pittsburgh Sleep Quality Index (PSQI) is a 19 item questionnaire that measures self-reported sleep quality and disturbances over the last 1 month time period. The questionnaire measures 7 components of sleep quality: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. A global PSQI score is obtained by summing the 7 component scores (range = 0-21). A PSQI global score > 5 indicates a poor sleeper.
Time Frame: baseline and 3 months after CPAP initiation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients in the Couple-oriented Intervention | Partners in the Couple-oriented Intervention | Patients in the Patient-oriented Intervention | Partners in the Patient-oriented Intervention | Patients in Usual Care | Partners in Usual Care
Number analyzed (Participants) | 5 | 5 | 6 | 6 | 9 | 9
units on a scale
  Baseline | 8.4 (2.5) | 7.0 (2.9) | 7.8 (3.1) | 7.2 (2.1) | 8.3 (4.5) | 9.9 (3.0)
  3 month follow-up | 5.0 (3.4) | 6.4 (5.0) | 5.8 (3.7) | 7.4 (3.7) | 6.1 (5.8) | 7.3 (2.8)
  Change from Baseline to 3 months | -4.3 (3.1) | -1.5 (3.5) | -2.0 (1.7) | -1.8 (2.2) | -2.2 (4.9) | -2.7 (4.4)
Statistical Analysis 1: Comparison: Patients in the Couple-oriented Intervention; Test type: Other; Effect size = -1.01
Statistical Analysis 2: Comparison: Patients in the Patient-oriented Intervention; Test type: Other; Effect size = -0.94
Statistical Analysis 3: Comparison: Patients in Usual Care; Test type: Other; Effect size = -0.40
Statistical Analysis 4: Comparison: Partners in the Couple-oriented Intervention; Test type: Other; Effect size = -0.31
Statistical Analysis 5: Comparison: Partners in the Patient-oriented Intervention; Test type: Other; Effect size = -0.65
Statistical Analysis 6: Comparison: Partners in Usual Care; Test type: Other; Effect size = -0.77

4. Secondary Outcome: Continuous Positive Airway Pressure (CPAP) Adherence
Description: Adherence will be measured as the amount of time that the CPAP machine is turned on and maintained at prescribed pressure. The latter number represents the amount of time power is on and the mask is positioned properly on the face. All patients will be using a CPAP machine with remote monitoring capabilities. Adherence reports are automatically uploaded to a secure data center daily. Adherence data can be accessed through the web-based patient compliance management system, EncoreAnywhere.
Time Frame: one week, one month, and 3 months after CPAP initiation
Measure: Mean (Standard Deviation); unit: hours of use
Arm/Group | Patients in the Couple-oriented Intervention | Patients in the Patient-oriented Intervention | Patients in Usual Care
Number analyzed (Participants) | 5 | 6 | 9
hours of use
  1 week | 5.6 (2.8) | 4.5 (2.6) | 5.8 (2.4)
  1 month | 6.1 (0.8) | 5.0 (2.9) | 5.1 (2.3)
  Change from 1 week to 1 month | 1.4 (1.9) | 0.5 (0.8) | -0.7 (0.7)
  3 months | 5.3 (2.9) | 4.5 (2.8) | 4.8 (2.4)
  Change from 1 month to 3 months | -1.6 (1.8) | -0.5 (0.6) | -0.3 (1.0)
Statistical Analysis 1: Comparison: Patients in the Couple-oriented Intervention; Test type: Other; Effect size = 0.52 — Comparing 1 week to 1 month
Statistical Analysis 2: Comparison: Patients in the Couple-oriented Intervention; Test type: Other; Effect size = -0.63 — Comparing 1 month and 3 months
Statistical Analysis 3: Comparison: Patients in the Patient-oriented Intervention; Test type: Other; Effect size = 0.50 — Comparing 1 week to 1 month
Statistical Analysis 4: Comparison: Patients in the Patient-oriented Intervention; Test type: Other; Effect size = -0.63 — Comparing 1 month to 3 months
Statistical Analysis 5: Comparison: Patients in Usual Care; Test type: Other; Effect size = -0.92 — Comparing 1 week to 1 month
Statistical Analysis 6: Comparison: Patients in Usual Care; Test type: Other; Effect size = -0.26 — Comparing 1 month to 3 months

ADVERSE EVENTS:
Arm/Group | Patients in the Couple-oriented Intervention | Partners in the Couple-oriented Intervention | Patients in the Patient-oriented Intervention | Partners in the Patient-oriented Intervention | Patients in Usual Care | Partners in Usual Care
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/10 | 0/10 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/10 | 0/10 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/10 | 0/10 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No